CLINICAL TRIAL: NCT05060887
Title: Phase 2a, Single Center, Randomized, Double-blind, Controlled Study to Evaluate the Immunogenicity and the Safety of One Single Administration of OVX836 Influenza Vaccine at Two Dose Levels (300μg and 480μg) Given Intramuscularly (IM), in Comparison to OVX836 Influenza Vaccine at 180μg and Placebo Given IM in Healthy Subjects Aged 18-55 Years and in Healthy Subjects Aged 65 Years and Older.
Brief Title: Immunogenicity and Safety of Three Dose Levels of OVX836 Candidate Vaccine Against Influenza in Healthy Volunteers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osivax (Industry)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OVX836-003
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized assignment to experimental vaccine (three dose levels) or placebo in a 1:1:1:1 ratio.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OVX836 - 180µg dose level (Experimental): Adjuvant-free recombinant influenza candidate vaccine based on the Nucleoprotein (NP) of the influenza virus. One single administration intramuscularly of a 180μg dose on Day 1.
  Interventions: Biological: OVX836-003
- OVX836 - 300µg dose level (Experimental): Adjuvant-free recombinant influenza candidate vaccine based on the Nucleoprotein (NP) of the influenza virus. One single administration intramuscularly of a 300μg dose on Day 1.
  Interventions: Biological: OVX836-003
- OVX836 - 480µg dose level (Experimental): Adjuvant-free recombinant influenza candidate vaccine based on the Nucleoprotein (NP) of the influenza virus. One single administration intramuscularly of a 480μg dose on Day 1.
  Interventions: Biological: OVX836-003
- Saline solution (B. Braun Ecoflac® Plus) (Placebo Comparator): Saline solution (NaCl 0.9%), B. Braun Ecoflac® Plus 50mL. One single administration intramuscularly of a 0.8mL dose on Day 1.
  Interventions: Biological: Saline solution

INTERVENTIONS:
Biological: OVX836-003 — One single administration intramuscularly at Day 1.
  Arms: OVX836 - 180µg dose level; OVX836 - 300µg dose level; OVX836 - 480µg dose level
Biological: Saline solution — One single administration intramuscularly at Day 1.
  Arms: Saline solution (B. Braun Ecoflac® Plus)

SUMMARY:
This Phase 2a clinical trial is designed to evaluate the immunogenicity and the safety of one administration of OVX836 influenza vaccine at different dose levels (180µg, 300μg and 480μg) in order to assess the dose response of the OVX836 influenza vaccine.

DETAILED DESCRIPTION:
This trial is a Phase 2a, randomized, double-blind, controlled study in 138 adult subjects to compare the immunogenicity and the safety of OVX836 influenza vaccine at two dose levels (300μg and 480μg) to lower dose level (180µg) and to placebo.

One single dose of OVX836 influenza vaccine (180µg or 300µg or 480µg) or of placebo will be administered intramuscularly in healthy subjects aged 18-55 years and in healthy subjects aged 65 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Healthy male or female subjects, as determined by medical history and medical examination.
3. Between the ages of 18 and 55 years, inclusive in the pilot phase and the first, younger age cohort; aged 65 years and older in the second, older age cohort..
4. Subject who has fully been vaccinated with licensed SARS-CoV-2 (COVID-19) vaccine(s) according to national recommendations for the corresponding population group.
5. Reliable and willing to make themselves available for the duration of the study, and willing and able to follow study procedures.
6. Ability and technical possibility for completing an e-diary and ePRO in the pilot phase and the first, younger age cohort; ability for completing a paper diary in the second, older age cohort.

Exclusion Criteria:

1. Subjects with a body mass index (BMI) ≤19 kg/m² or ≥35 kg/m² on the day of vaccination.
2. In the pilot phase and the first younger age cohort only: Previous influenza vaccination within 6 months before the day of vaccination or planned to receive during the study duration.
3. Any known or suspected immunodeficient conditions.
4. Past or current history of significant autoimmune diseases, as judged by the Investigator.
5. Current history of uncontrolled medical illness such as diabetes, hypertension, heart, renal or hepatic diseases.
6. Known or suspected infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
7. Female subjects: pregnant, breast-feeding or of childbearing potential without appropriate contraceptive methods in place for 2 months before enrolment, or with positive pregnancy test on the day of vaccination. Appropriate contraceptive methods are to be maintained until the end of the trial. Appropriate contraceptive methods are defined by the Clinical Trial Facilitation Group [CTFG] as follow: "Contraceptive methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include: combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable intrauterine device, intrauterine hormonereleasing system), bilateral tubal occlusion, vasectomized partner and/or sexual abstinence (refraining from heterosexual intercourse)."
8. Having received another vaccination within 3 months prior to the day of study vaccination for live attenuated vaccines, or within 1 month prior to the day of study vaccination for inactivated vaccines, except COVID-19 vaccine.
9. Planning to receive other vaccines during the first 28 days following the study vaccine administration, except COVID-19 vaccine.
10. Administration of any investigational or non-registered drug or vaccine within 3 months prior to the administration of study vaccines, or planned administration of any such product during the whole study period.
11. History of receiving blood, blood components or immunoglobulins within 3 months prior to the day of vaccination, or planned to receive such product during the whole study period.
12. Presence of an acute febrile illness on the day of vaccination (oral temperature >38.0°C, temporary exclusion criterion).
13. Past or current history of any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
14. Behavioral or cognitive impairment, or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.
15. Past (stopped less than 6 months before enrolment) or current history of alcohol or drug abuse, or current smoking habit above 10 cigarettes per day, or current vaping.
16. Treatment that can affect immune response such as systemic or high dose inhaled corticosteroids (>800μg/day beclomethasone or equivalent; occasional inhaled corticosteroids for asthma therapy are allowed), radiation treatment, cytotoxic drugs, or current or recent (within 30 days before study entry) chronic or prolonged (>10 days) use of systemic non-steroidal anti-inflammatory drugs, interferon, immunomodulators, allergy shots, as judged by the Investigator.
17. History of severe allergic reactions and/or anaphylaxis, or serious adverse reactions to vaccines or allergy to kanamycin.
18. Any contraindication to IM administration, as judged by the Investigator.
19. Individuals with history of any illness that, in the opinion of the Investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
20. Sponsor employees or Investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted, including children of newly composed families.
21. Previous administration with OVX836 candidate vaccine.
22. Having received a COVID-19 vaccination within 2 weeks prior to the day of study vaccination.
23. Planning to receive COVID-19 vaccine during the first week (within 7 days) following the study vaccine administration. An interval of preferably 14 days is recommended. If for scheduling reasons, COVID-19 vaccine has to be given on Day 8, the vaccination should be administered after completion of the study procedures.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Change of NP-specific T-cell frequencies in peripheral blood, measured by IFNγ ELISPOT, at Day 8 versus pre-injection baseline (Day 1). | at Day 8 versus pre-injection baseline (Day 1)
Proportion of subjects reporting solicited local (Injection site redness, Injection site swelling, Injection site pain) and systemic symptoms (Fatigue, Headache, Arthralgia, Malaise, Myalgia, Fever) | during 7 days after vaccine administration
Proportion of subjects reporting unsolicited Adverse Events | during 29 days after vaccine administration
Proportion of subjects with Influenza-Like-Illness cases associated with laboratory-confirmed influenza | during the whole study duration, 180 days
Severity scores of Influenza-Like-Illness cases (as per Flu-PRO® questionnaire) | during the whole study duration, 180 days
Proportion of subjects reporting Serious Adverse Events | during the whole study duration, 180 days

SECONDARY OUTCOMES:
NP-specific IFNγ T-cell activity measured by ELISPOT | at Day 8 and Day 180 versus pre-injection baseline (Day 1)
NP-specific CD4+ and CD8+T-cell frequencies measured by flow cytometry (on PBMCs) as expressing IL-2, TNFα and/or IFNγ upon in vitro stimulation at Day 1 (pre-injection baseline), Day 8 and Day 180. | at Day 1 (pre-injection baseline), Day 8 and Day 180
Anti-NP Immunoglobulin G (IgG) titers by ELISA at each time point | at Day 1 (pre-injection baseline), Day 8, Day 29 and Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Leroux-Roels, MD, PhD, Principal Investigator — Centre for Vaccinology (CEVAC), Ghent University Hospital
Locations (1):
- Centre for Vaccinology (CEVAC), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leroux-Roels I, Willems P, Waerlop G, Janssens Y, Tourneur J, De Boever F, Bruhwyler J, Alhatemi A, Jacobs B, Nicolas F, Leroux-Roels G, Le Vert A. Immunogenicity, safety, and preliminary efficacy evaluation of OVX836, a nucleoprotein-based universal influenza A vaccine candidate: a randomised, double-blind, placebo-controlled, phase 2a trial. Lancet Infect Dis. 2023 Dec;23(12):1360-1369. doi: 10.1016/S1473-3099(23)00351-1. Epub 2023 Jul 27. PMID 37517422
- See also: Related Info — https://doi.org/10.1016/S1473-3099(23)00351-1